CLINICAL TRIAL: NCT01163357
Title: Phase I Study of Bortezomib With or Without Total Marrow Irradiation (TMI) Using Intensity Modulated Radiation Therapy (IMRT) in Combination With Fludarabine (FLU) and Melphalan (MEL) as a Preparative Regimen for Allogeneic Hematopoietic Stem Cell (HSC) Transplantation in Patients With High Risk Multiple Myeloma
Brief Title: Bortezomib, Total Marrow Irradiation, Fludarabine Phosphate, and Melphalan in Treating Patients Undergoing Donor Peripheral Blood Stem Cell Transplant For High-Risk Stage I or II Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09171; NCI-2010-01610 (Other: NCI CTRP)
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Autologous Hematopoietic Stem Cell Transplant Recipient; Loss of Chromosome 17p; Plasma Cell Leukemia; Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Chromosome 17 deletion; Leukemia, Plasma Cell; Multiple Myeloma | interventions — Bortezomib; fludarabine phosphate; Melphalan; Tacrolimus; Sirolimus; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (bortezomib, fludarabine phosphate, TMI, melphalan) (Experimental): Patients receive fludarabine phosphate IV on days -9 to -5 and melphalan IV on day -4. Patients also undergo TMI BID on days -9 to -7. If no DLT is observed in the first cohort, bortezomib IV will be added on days -6 and -3 for subsequent cohorts.
  Interventions: Drug: bortezomib; Drug: fludarabine phosphate; Other: melphalan; Radiation: total marrow irradiation; Drug: tacrolimus; Drug: sirolimus; Procedure: peripheral blood stem cell transplantation; Other: laboratory biomarker analysis
- Group II (bortezomib, fludarabine phosphate, melphalan (Experimental): Patients receive fludarabine phosphate IV and melphalan IV as in Stratum I. Patients also receive bortezomib IV on days -6, -3, 1, and 4.
  Interventions: Drug: bortezomib; Drug: fludarabine phosphate; Other: melphalan; Drug: tacrolimus; Drug: sirolimus; Procedure: peripheral blood stem cell transplantation; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; PS-341; VELCADE
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Other: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin; Melfalan
Radiation: total marrow irradiation — Undergo TMI
  Arms: Group I (bortezomib, fludarabine phosphate, TMI, melphalan)
Drug: tacrolimus — Given IV and orally
  Other Names: Advagraf; FK 506; Prograf; Protopic
Drug: sirolimus — Given orally
  Other Names: AY 22989; RAPA; Rapamune; rapamycin; SILA 9268A; SLM
Procedure: peripheral blood stem cell transplantation — Undergo allogeneic PBSC transplant
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving chemotherapy drugs, such as fludarabine phosphate and melphalan, and total marrow irradiation before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets.

PURPOSE: This phase I trial is studying the side effects and best dose of bortezomib when given together with fludarabine phosphate and melphalan with or without total marrow irradiation in treating patients undergoing donor peripheral blood stem cell transplant for high-risk stage I or II multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of escalating doses of bortezomib with or without total marrow irradiation (TMI) at a fixed dose of 900 cGy in combination with fludarabine (FLU) and melphalan (MEL) as preparative regimen for allogeneic hematopoietic stem cell transplant in patients with high risk multiple myeloma who have human leukocyte antigen (HLA) matched donor (sibling or matched unrelated donor).

II. To describe toxicities, maximum tolerated dose (MTD) and dose limiting toxicities (DLT) of this preparative regimen.

SECONDARY OBJECTIVES:

I. To evaluate the frequency of clinical response, i.e., complete response [CR], partial response [PR], very good partial response [VGPR]) at 6 month and 1 year post transplant.

II. To evaluate the frequency of primary and secondary engraftment failure.

III. To evaluate the time to neutrophil and platelet engraftment.

IV. To evaluate the incidence of acute and chronic graft-versus-host disease (GVHD).

V. To evaluate progression-free survival.

VI. To evaluate overall survival.

VII. To evaluate minimal residual disease (MRD) at 6 months and 1 year post transplant by flow cytometry in the bone marrow.

OUTLINE: This is a dose-escalation study of bortezomib. Patients are assigned to 1 of 2 treatment groups. GROUP I (patients eligible for TMI): Patients receive fludarabine phosphate intravenously (IV) on days -9 to -5 and melphalan IV on day -4. Patients also undergo TMI twice daily (BID) on days -9 to -7. If no DLT is observed in the first cohort, bortezomib IV will be added on days -6 and -3 for subsequent cohorts. GROUP II (patients ineligible for TMI): Patients receive fludarabine phosphate IV and melphalan IV as in Group I. Patients also receive bortezomib IV on days -6, -3, 1, and 4.

TRANSPLANT: All patients undergo allogeneic peripheral blood stem cell (PBSC) transplant on day 0.

GVHD PROPHYLAXIS: All patients receive tacrolimus IV or orally (PO) and sirolimus PO beginning on day -3.

After completion of study treatment, patients are followed up at day 100, 6 months, and then annually thereafter for up to 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Recipient must have signed a voluntary, informed consent in accordance with institutional and federal guidelines
* Recipients must have histopathologically confirmed diagnosis of multiple myeloma
* Age:

  * Stratum I (TMI containing arm): 18-60 years of age
  * Stratum II (non TMI arm): 18-70 years of age
* Patients with primary progressive disease on induction therapy with new targeted therapies
* Relapsed/refractory disease on new targeted therapies, i.e. thalidomide, lenalidomide, bortezomib, or other new novel agents such as carfilzomib, pomalidomide
* Patients with relapsed multiple myeloma following previous autologous stem cell transplant
* Plasma cell leukemia at diagnosis
* High-risk patients with presence of chromosome 17p deletion (> 60%) in the bone marrow by fluorescence in situ hybridization (FISH); patients are not required to have prior autologous stem cell transplant
* Able to lie supine for approximately 60 minutes, the anticipated duration of each treatment session
* Performance status evaluated by Eastern Cooperative Oncology Group (ECOG) or Karnofsky Performance Scales (KPS) patients must have a score of 0-II (ECOG) or >= 70% (KPS)
* Cardiac ejection fraction >= 50% by multiple gate acquisition (MUGA) scan and/or by echocardiogram
* Forced expiratory volume in one second (FEV1) >= 50%
* Diffusing lung capacity for carbon monoxide (DLCO) >= 50%
* Creatinine clearance or glomerular filtration rate (GFR) >= 60 ml/min
* Serum bilirubin =< 2.0 mg/dl
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) =< 2.5 times the institutional upper limits of normal
* Pre-treatment tests must be performed within 30 days prior to enrollment
* No other medical and or psychosocial problems, which in the opinion of the primary physician or principal investigator would place the patient at unacceptable risk from this regimen
* Patients with no previous radiation or up to a maximum 2000 cGy to non thoracic-spine and rib bone lesions or < 20% of bone marrow are eligible for TMI conditioning regimen
* Patients with previous history of irradiation at any dose to thoracic-spine, ribs or >= 20% of bone marrow cannot undergo TMI and will be eligible for bortezomib, fludarabine, and melphalan regimen

Stratum II); patients can be enrolled on stratum II at their physician's discretion or if patients decline radiation therapy

DONOR: Any matched sibling donor (matched at HLA A, B, C by intermediate resolution typing and HLA-DRB1 by high resolution typing), or unmatched unrelated donor (matched at HLA A, B, C, DRB1 by high resolution typing) will be considered a suitable donor

Exclusion Criteria:

* Patients with peripheral neuropathy greater than grade II
* Major medical or psychiatric disorders that would seriously compromise patient tolerance of this regimen
* Human immunodeficiency virus (HIV) infection, active hepatitis B or C infection, or evidence of liver cirrhosis
* Active viral, bacterial or fungal infection unless adequately treated. For fungal infection, patient should have completed full course of antifungal therapy with resolution of infection.
* Patients with radiographic changes including pulmonary disease, including but not limited to: pulmonary nodules, infiltrates, pleural effusion are excluded unless cleared by pulmonary biopsy showing no evidence for pulmonary infection
* Patients with renal insufficiency or cr clearance < 60 ml/min

DONOR: Donors will be excluded if for medical or psychological reasons they are unable to tolerate the procedure of peripheral stem cell donation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-01-28 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of bortezomib as defined as the highest dose tested in which none or only one patient experiences dose limiting toxicity attributable to the study regimen | 6 weeks post transplant
  Assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Dose-limiting toxicity will be defined using Bearman Scale for events that occur.
Feasibility of escalating doses of bortezomib with or without TMI in combination with FLU and MEL as preparative regimen for allogeneic hematopoietic stem cell transplant in patients with high risk multiple myeloma | 5 years post transplant

SECONDARY OUTCOMES:
Frequency of clinical response (i.e., complete, partial, or very good partial response) | At 6 months and 1 year post transplant
  Response is evaluated based on a new International myeloma working group uniform response criteria.
Frequency of primary and secondary engraftment failure | 6 weeks post transplant and 4 years post transplant
Time to neutrophil and platelet engraftment | 100 days post transplant
Progression-free survival | 4 years post transplant
  Time from day 0 of transplant to the first observation or relapse or death due to any cause, assessed up to 4 years
Incidence of acute and chronic graft-versus-host disease | At 6 months and 1 year post transplant up to 4 years post transplant
Overall survival | 4 years post transplant
  Time from first day of treatment to time of death due to any cause, assessed up to 4 years
Minimal residue disease | At 6 months and 1 year post transplant
  Assessed by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Firoozeh Sahebi, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States